CLINICAL TRIAL: NCT04226326
Title: Investigating the Utility of Remote Index of Microvascular Resistance in Patients With Chronic Total Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB19-0654
Record Dates: First submitted 2019-12-18; First posted 2020-01-13 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Chronic Total Occlusion
Keywords: Microvascular Resistance; Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with Chronic Total Occlusion (CTO) (Other): All subjects in this study have been scheduled for a clinically-indicated cardiac catheterization.
  Interventions: Other: Directly measure microvascular function using direct coronary flow measurements

INTERVENTIONS:
Other: Directly measure microvascular function using direct coronary flow measurements — The study will enroll subjects who have been scheduled for a clinically-indicated cardiac catheterization, and will evaluate coronary microvascular function in all subjects meeting inclusion criteria with a coronary flow wire. Evaluation of coronary microvascular function may be performed using indirect methods, however the rationale behind the present study is to directly measure microvascular function using direct coronary flow measurements, since the subjects in the study are to undergo a clinically-indicated cardiac catheterization. The overall purpose of the study is to define the presence and severity of coronary microvascular dysfunction subjects with CTO.

SUMMARY:
This is prospective cohort study in subjects with a planned percutaneous coronary intervention (PCI) of their chronic total occlusion (CTO). The study will enroll subjects who have been scheduled for a clinically-indicated cardiac catheterization, and will evaluate coronary microvascular function in all subjects meeting inclusion criteria with a coronary flow wire. Evaluation of coronary microvascular function may be performed using indirect methods, however the rationale behind the present study is to directly measure microvascular function using direct coronary flow measurements, since the subjects in the study are to undergo a clinically-indicated cardiac catheterization. The overall purpose of the study is to define the presence and severity of coronary microvascular dysfunction subjects with CTO. The study is designed to enroll 50 subjects with CTO in the span of 3 years. There will be a 6-month assessment of the outcomes of death and cardiovascular death. As the study includes FDA approved tests, there will be no safety endpoint per se, however there will be a mechanism for monitoring adverse events as will be described in detail.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 21 years
* seen at University of Chicago Medical center with a planned PCI of a single CTO vessel
* must have either stable angina or angina equivalent
* must have a CTO with a clear donor vessel supplying most of the collaterals.

Exclusion Criteria:

* subjects with a pacemaker or implantable cardioverter defibrillator
* contraindication to cardiac MRI, adenosine, heparin, or nitroglycerin
* cardiac transplantation
* Estimated glomerular filtration rate (eGFR) ≤ 30 mL/min/1.73m2, given the risk of contrast-induced nephropathy (CIN) and nephrogenic systemic fibrosis (NSF) associated with iodinated and gadolinium-based contrast agents, respectively, in patients with significant renal dysfunction
* Women who may potentially be pregnant will receive a pregnancy test and be excluded if pregnant
* Vulnerable populations such as children, college students, prisoners, non-English speakers, and those with diminished decision-making capacity
* Inability or refusal to consent for the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Baseline myocardial quality of the CTO-supplied vascular bed. | Day of procedure
  Characterize the microvascular resistance of the donor vessel to 50 CTOs as it relates to vascular bed quality of the CTO-supplied territory. Scaled from 0-102, with 102 being worse than 0.
  1. Baseline myocardial quality
IMR of opened CTO vessel | 6 months
  Following CTO PCI, IMR of the opened vessel will be measured. Scale is linear and 1-100 units, higher numbers being worse outcome.
  3) Change in SAQ from baseline to 6 months
Change in exercise time on Bruce protocol baseline | 6 months
  Change in exercise time from baseline to 6 months post-PCI will be measured. Scale is linear and measured in seconds (can be a negative number), with higher numbers indicating a favorable outcome.
Change in SAQ from baseline to 6 months | 6 months
  Change in Seattle Angina Questionnaire (SAQ) from baseline to 6 months post-PCI will be measured. Scale is linear and 0-100 units, with higher numbers indicating a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John Blair, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Ramunddal T, Hoebers LP, Henriques JP, Dworeck C, Angeras O, Odenstedt J, Ioanes D, Olivecrona G, Harnek J, Jensen U, Aasa M, Jussila R, James S, Lagerqvist B, Matejka G, Albertsson P, Omerovic E. Chronic total occlusions in Sweden--a report from the Swedish Coronary Angiography and Angioplasty Registry (SCAAR). PLoS One. 2014 Aug 12;9(8):e103850. doi: 10.1371/journal.pone.0103850. eCollection 2014. PMID 25117457
- [Background] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Background] Claessen BE, van der Schaaf RJ, Verouden NJ, Stegenga NK, Engstrom AE, Sjauw KD, Kikkert WJ, Vis MM, Baan J Jr, Koch KT, de Winter RJ, Tijssen JG, Piek JJ, Henriques JP. Evaluation of the effect of a concurrent chronic total occlusion on long-term mortality and left ventricular function in patients after primary percutaneous coronary intervention. JACC Cardiovasc Interv. 2009 Nov;2(11):1128-34. doi: 10.1016/j.jcin.2009.08.024. PMID 19926056
- [Background] Puma JA, Sketch MH Jr, Tcheng JE, Gardner LH, Nelson CL, Phillips HR, Stack RS, Califf RM. The natural history of single-vessel chronic coronary occlusion: a 25-year experience. Am Heart J. 1997 Apr;133(4):393-9. doi: 10.1016/s0002-8703(97)70179-0. PMID 9124159
- [Background] Farooq V, Serruys PW, Garcia-Garcia HM, Zhang Y, Bourantas CV, Holmes DR, Mack M, Feldman T, Morice MC, Stahle E, James S, Colombo A, Diletti R, Papafaklis MI, de Vries T, Morel MA, van Es GA, Mohr FW, Dawkins KD, Kappetein AP, Sianos G, Boersma E. The negative impact of incomplete angiographic revascularization on clinical outcomes and its association with total occlusions: the SYNTAX (Synergy Between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery) trial. J Am Coll Cardiol. 2013 Jan 22;61(3):282-94. doi: 10.1016/j.jacc.2012.10.017. Epub 2012 Dec 19. PMID 23265332
- [Background] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Background] Bagnall A, Spyridopoulos I. The evidence base for revascularisation of chronic total occlusions. Curr Cardiol Rev. 2014 May;10(2):88-98. doi: 10.2174/1573403x10666140331125659. PMID 24694105
- [Background] Brilakis ES, Banerjee S, Karmpaliotis D, Lombardi WL, Tsai TT, Shunk KA, Kennedy KF, Spertus JA, Holmes DR Jr, Grantham JA. Procedural outcomes of chronic total occlusion percutaneous coronary intervention: a report from the NCDR (National Cardiovascular Data Registry). JACC Cardiovasc Interv. 2015 Feb;8(2):245-253. doi: 10.1016/j.jcin.2014.08.014. PMID 25700746
- [Background] Henriques JP, Hoebers LP, Ramunddal T, Laanmets P, Eriksen E, Bax M, Ioanes D, Suttorp MJ, Strauss BH, Barbato E, Nijveldt R, van Rossum AC, Marques KM, Elias J, van Dongen IM, Claessen BE, Tijssen JG, van der Schaaf RJ; EXPLORE Trial Investigators. Percutaneous Intervention for Concurrent Chronic Total Occlusions in Patients With STEMI: The EXPLORE Trial. J Am Coll Cardiol. 2016 Oct 11;68(15):1622-1632. doi: 10.1016/j.jacc.2016.07.744. PMID 27712774